CLINICAL TRIAL: NCT05638399
Title: Denosumab vs Zoledronate Efficacy in Osteopenic Patients With Lumbar Degenerative Disease After Lumbar Fusion Surgery
Brief Title: Denosumab vs Zoledronate After Lumbar Fusion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShenzhenPH spine06
Record Dates: First submitted 2022-11-25; First posted 2022-12-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Osteopenia; Lumbar Spondylolisthesis
MeSH Terms: conditions — Bone Diseases, Metabolic; Spondylolisthesis | interventions — Denosumab; Injections, Subcutaneous; Zoledronic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Experimental): denosumab (60 mg subcutaneously, per 6 month)
  Interventions: Drug: Denosumab 60 mg/ml [Prolia]
- zoledronate (Active Comparator): zoledronate (5mg, intravenous infusion once a year)
  Interventions: Drug: Zoledronate

INTERVENTIONS:
Drug: Denosumab 60 mg/ml [Prolia] — 60 mg subcutaneously per 6 month
  Other Names: Denosumab 6 month/subcutaneous
  Arms: Denosumab
Drug: Zoledronate — 5mg, intravenous infusion once a year
  Other Names: Zoledronic acid
  Arms: zoledronate

SUMMARY:
The aim of the study was to compare denosumab and zoledronate efficacy in bone mass, bone turnover markers (BTMs), Visual Analogue Scale (VAS) for leg and back, EuroQol Five-Dimension (EQ-5D) scores, Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 (QUALEFFO-31) scores, and Roland-Morris Disability Functioning Questionnaire (RMDQ) scores, secondary fracture, complications and adverse events after lumbar fusion.

DETAILED DESCRIPTION:
Lumbar degenerative disease including spinal stenosis and lumbar spondylolisthesis were the most common reason lead to older patients disability, which was the main indication for older patients to perform lumbar fusion surgery. For patients with lumbar degenerative disease older than 50 years old, a proportion of patients had osteoporosis. The trial aims to investigate whether denosumab versus zoledronate acid in osteopenic patients with lumbar fusion surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 40 to 85 years

  * who diagnosed with lumbar spinal stenosis or lumbar spondylolisthesis
  * osteopenia with BMD T score between -1 and -2.5 via dual energy X-ray
  * low back pain or leg numbness or weakness
  * MRI demonstrated signs of nerve compression
  * patients with one or two level symptoms.

Exclusion Criteria:

* cauda equina syndrome

  * progressive neurologic deficit
  * history of cancer
  * scoliosis greater than 15°
  * back open surgery history
  * have contraindications for surgery
  * who had anti-osteoporosis medication within 6 weeks

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-02-26 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Lumbar bone mineral density(BMD) | up to 12 months
  Lumbar vertebral (L1 to L4, except the surgery segment) BMD were determined at baseline, 6 and 12 months via dual energy X-ray
Total hip BMD | up to 12 months
  Total hip BMD were determined at baseline, 6 and 12 months via dual-energy X-ray
Femoral neck BMD | up to 12 months
  Femoral neck BMD were determined at baseline, 6 and 12 month via dual-energy X-ray
Procollagen type 1 n-terminal propeptide (P1NP) | up to 12 months
  Bone formation marker, P1NP were determined at baseline, 6 and 12 months after surgery
C-terminal cross-linked type 1 collagen terminal peptide (CTX) | up to 12 months
  Bone resorption marker, CTX were determined at baseline, 6 and 12 months after surgery
Visual analog scale (VAS) back | up to 12 months
  The VAS score for back pain were determined at baseline, 6 and 12 month. Use a ruler about 10cm long, one side is marked with "0" and the other "10" respectively. A score of 0 indicates no pain, 10 indicates the most unbearable pain.

SECONDARY OUTCOMES:
The Roland-Morris Disability Questionnaire | up to 12 month
  The Roland-Morris Disability Questionnaire is scored by 24 adding up the number of items checked "yes" on different low back pain-related daily activity disabilities. Total scores range from 0 to 24, with higher scores 24 indicating a higher level of disability related to low back pain and lowest 0 represents no back pain.
The QUALEFFO-31 Questionnaire | up to 12 month
  The Quality of Life Questionnaire of the European Foundation for Osteoporosis-31 (QUALEFFO-31), which contains three domains including pain, physical function, and mental function. This scale is assessed on a scale of 0 to 100, with 0 indicating the highest QoL and 100 the lowest.
The EQ-5D Questionnaire | up to 12 month
  The EuroQol five-dimension (EQ-5D) questionnaire evaluates health status consisting five dimensions: mobility, selfcare, performance of usual activities, pain or discomfort, and anxiety or depression. After conversion, the index was between 0 and 1.0 (minimum score: 0, indicating worst health state; full score:1.0, indicating full health).
New fracture rate | up to 12 month
  New fracture rate containing vertebral fracture and non-vertebral fracture was assessed at 12 month after surgery. The lowest score was 0, the highest score was 100%. The lower score 0 represents no secondary fracture.
Complications | up to 12 month
  Complications including cage subsidence, pedicle screw loosening, infection, peripheral nerve injury, and recurrent symptoms were assessed.
Adverse events | up to 12 month
  The main adverse events including deep venous thrombosis, pneumonia, acute renal failure, pulmonary embolism, myocardial infarction, influenza, transfer to intensive care unit, joint pain, headache, nausea, osteonecrosis of the jaw, atypical femoral fracture and rash.

CONTACTS AND LOCATIONS:
Overall Officials: Songlin Peng, Doctor, Study Chair — Shenzhen People's Hospital
Locations (1):
- ShenzhenPH, Shenzhen, Guangdong, China